CLINICAL TRIAL: NCT01405976
Title: Mid-and Long-term Efficacy of Ventilation Non-invasive and Continuos Positive Airway Pressure in Obesity Hypoventilation Syndrome
Brief Title: Alternative of Treatment in Obesity Hypoventilation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI080346
Record Dates: First submitted 2008-07-03; First posted 2011-07-29 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-01

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: sleep apneas; noninvasive ventilation; CPAP
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea Syndromes | interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): NIV for severe OSA group
  Interventions: Device: life style modification, noninvasive ventilation, CPAP
- 2 (Active Comparator): CPAP for severe OSA group
  Interventions: Device: life style modification, noninvasive ventilation, CPAP
- 3 (Active Comparator): Life stile modification for severe OSA group
  Interventions: Device: life style modification, noninvasive ventilation, CPAP
- 4 (Active Comparator): NIV for non-severe OSA group
  Interventions: Device: life style modification, noninvasive ventilation, CPAP
- 5 (Active Comparator): Life stile modification for non-severe OSA group
  Interventions: Device: life style modification, noninvasive ventilation, CPAP

INTERVENTIONS:
Device: life style modification, noninvasive ventilation, CPAP — life style modification, noninvasive ventilation, CPAP

SUMMARY:
Primary objectives: evaluate the efficacy of noninvasive ventilation (NIV) treatment versus continuous positive airway pressure (CPAP) and life style modification treatment in Obesity Hypoventilation Syndrome (OHS), with PCO2 (first phase) and days of hospitalization (second phase) analyzed as a primary variables and percentage of dropouts for medical reasons and mortality as operative variables. As secondary variables: Measure functional and clinical improvement during sleep and wakefulness, quality of life, echocardiography and the incidence and blood pressure and evolution of cardiovascular events. Objectives secondaries:role of apneogenic sleep events on molecular inflammation, endothelial damage and the genesis of diurnal hypercapnia. Methods:prospective, randomized controlled trial. Patients with OHS will be divided initially into two groups based on their apnea-hypopnea index (AHI) score, >=30 and < 30, using conventional polysomnography. The AHI >=30 group will be randomized to CPAP, NIV or life style modification treatments. The AHI <=30 groups will be randomized to NIV or life style modification treatments. Treatment efficacy at the medium- and long-term will be analyzed by comparing groups. The role of apneic events and leptin in the genesis of daytime alveolar hypoventilation will be analyzed by comparing the daytime PCO2/AHI coefficient between responders and non-responders to CPAP treatment, and the evolution of leptin levels in the four branches of the study. The role of apneic events in metabolic and biochemical alterations and endothelial dysfunction will be analyzed by comparing basal and post-treatment levels of related substances between groups, with and without significant AHI.

DETAILED DESCRIPTION:
The AHI >=30 group will be analyzed to CPAP, NIV or life style modification treatments for two mouths.Once an evaluation is done during this period, the life style modification treatment will be randomized with the NIV/CPAP treatment for a continuation of three years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 80 years old.
* Absence of moderate or severe chronic obstructive pulmonary disease (COPD).
* Absence of neuromuscular, chest wall or metabolic disease which cause daytime hypercapnia.
* Absence of narcolepsy or restless legs syndrome
* Exceed correctly treatment of at least 30 minutes with CPAP/NIV at wakefulness.

Exclusion Criteria:

* Psychophysical incapacity to answer questionnaires.
* Patients who are not able to be evaluated by means of quality of life questionnaires for suffering restrictive chronic disease previously diagnosed (neoplasy, chronic pain of any origin, renal failure, severe chronic obstructive pulmonary disease and any other restrictive chronic disease).
* Subjects with important chronic nasal obstruction that prevents from using CPAP/NIV.
* Informed consent not obtained.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Days of hospitalization | at least three years
  Days of hospitalization
PaCO2 | at the end of first two months
  PaCO2

SECONDARY OUTCOMES:
Number of Dropouts for Medical reasons and mortality | at least three years
  Number of Dropouts for Medical reasons and mortality
quality of life | two months and three years
  quality of life
respiratory function | two months and three years
  respiratory function
polysomnographic parameters | two months
  polysomnographic parameters
molecular inflammation and endothelial dysfunction | two months and three years
  molecular inflammation and endothelial dysfunction
echocardiographic parameters | two months and three years
  echocardiographic parameters
Blood pressure and new cardiovascular events | three years
  Blood pressure and new cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Masa, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Hospital San Pedro de Alcántara. Servicio Extremeño de Salud, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masa JF, Benitez ID, Javaheri S, Mogollon MV, Sanchez-Quiroga MA, de Terreros FJG, Corral J, Gallego R, Romero A, Caballero-Eraso C, Ordax-Carbajo E, Troncoso MF, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Barbe F, Mokhlesi B; Spanish Sleep Network. Risk factors associated with pulmonary hypertension in obesity hypoventilation syndrome. J Clin Sleep Med. 2022 Apr 1;18(4):983-992. doi: 10.5664/jcsm.9760. PMID 34755598
- [Derived] Masa JF, Benitez I, Sanchez-Quiroga MA, Gomez de Terreros FJ, Corral J, Romero A, Caballero-Eraso C, Alonso-Alvarez ML, Ordax-Carbajo E, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Vazquez-Polo FJ, Negrin MA, Martel-Escobar M, Barbe F, Mokhlesi B; Spanish Sleep Network. Long-term Noninvasive Ventilation in Obesity Hypoventilation Syndrome Without Severe OSA: The Pickwick Randomized Controlled Trial. Chest. 2020 Sep;158(3):1176-1186. doi: 10.1016/j.chest.2020.03.068. Epub 2020 Apr 25. PMID 32343963
- [Derived] Masa JF, Mokhlesi B, Benitez I, Gomez de Terreros Caro FJ, Sanchez-Quiroga MA, Romero A, Caballero C, Alonso-Alvarez ML, Ordax-Carbajo E, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Vazquez-Polo FJ, Negrin MA, Martel-Escobar M, Barbe F, Corral-Penafiel J; Spanish Sleep Network. Cost-effectiveness of positive airway pressure modalities in obesity hypoventilation syndrome with severe obstructive sleep apnoea. Thorax. 2020 Jun;75(6):459-467. doi: 10.1136/thoraxjnl-2019-213622. Epub 2020 Mar 26. PMID 32217780
- [Derived] Masa JF, Mokhlesi B, Benitez I, Mogollon MV, Gomez de Terreros FJ, Sanchez-Quiroga MA, Romero A, Caballero-Eraso C, Alonso-Alvarez ML, Ordax-Carbajo E, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Vazquez-Polo FJ, Negrin MA, Martel-Escobar M, Barbe F, Corral J; Spanish Sleep Network. Echocardiographic Changes with Positive Airway Pressure Therapy in Obesity Hypoventilation Syndrome. Long-Term Pickwick Randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2020 Mar 1;201(5):586-597. doi: 10.1164/rccm.201906-1122OC. PMID 31682462
- [Derived] Masa JF, Mokhlesi B, Benitez I, Gomez de Terreros FJ, Sanchez-Quiroga MA, Romero A, Caballero-Eraso C, Teran-Santos J, Alonso-Alvarez ML, Troncoso MF, Gonzalez M, Lopez-Martin S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Barca J, Vazquez-Polo FJ, Negrin MA, Martel-Escobar M, Barbe F, Corral J; Spanish Sleep Network. Long-term clinical effectiveness of continuous positive airway pressure therapy versus non-invasive ventilation therapy in patients with obesity hypoventilation syndrome: a multicentre, open-label, randomised controlled trial. Lancet. 2019 Apr 27;393(10182):1721-1732. doi: 10.1016/S0140-6736(18)32978-7. Epub 2019 Mar 29. PMID 30935737
- [Derived] Corral J, Mogollon MV, Sanchez-Quiroga MA, Gomez de Terreros J, Romero A, Caballero C, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martinez S, de Lucas P, Marin JM, Romero O, Diaz-Cambriles T, Chiner E, Egea C, Lang RM, Mokhlesi B, Masa JF; Spanish Sleep Network. Echocardiographic changes with non-invasive ventilation and CPAP in obesity hypoventilation syndrome. Thorax. 2018 Apr;73(4):361-368. doi: 10.1136/thoraxjnl-2017-210642. Epub 2017 Nov 16. PMID 29146865
- [Derived] Masa JF, Corral J, Romero A, Caballero C, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martinez S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Merchan M, Egea C, Obeso A, Mokhlesi B; Spanish Sleep Network. The Effect of Supplemental Oxygen in Obesity Hypoventilation Syndrome. J Clin Sleep Med. 2016 Oct 15;12(10):1379-1388. doi: 10.5664/jcsm.6194. PMID 27568890
- [Derived] Masa JF, Corral J, Caballero C, Barrot E, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Egea C, Miranda E, Mokhlesi B; Spanish Sleep Network; Garcia-Ledesma E, Sanchez-Quiroga MA, Ordax E, Gonzalez-Mangado N, Troncoso MF, Martinez-Martinez MA, Cantalejo O, Ojeda E, Carrizo SJ, Gallego B, Pallero M, Ramon MA, Diaz-de-Atauri J, Munoz-Mendez J, Senent C, Sancho-Chust JN, Ribas-Solis FJ, Romero A, Benitez JM, Sanchez-Gomez J, Golpe R, Santiago-Recuerda A, Gomez S, Bengoa M. Non-invasive ventilation in obesity hypoventilation syndrome without severe obstructive sleep apnoea. Thorax. 2016 Oct;71(10):899-906. doi: 10.1136/thoraxjnl-2016-208501. Epub 2016 Jul 12. PMID 27406165
- [Derived] Masa JF, Corral J, Romero A, Caballero C, Teran-Santos J, Alonso-Alvarez ML, Gomez-Garcia T, Gonzalez M, Lopez-Martin S, De Lucas P, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Merchan M, Egea C, Obeso A, Mokhlesi B; Spanish Sleep Network( *). Protective Cardiovascular Effect of Sleep Apnea Severity in Obesity Hypoventilation Syndrome. Chest. 2016 Jul;150(1):68-79. doi: 10.1016/j.chest.2016.02.647. Epub 2016 Feb 27. PMID 26923627
- [Derived] Masa JF, Corral J, Alonso ML, Ordax E, Troncoso MF, Gonzalez M, Lopez-Martinez S, Marin JM, Marti S, Diaz-Cambriles T, Chiner E, Aizpuru F, Egea C; Spanish Sleep Network. Efficacy of Different Treatment Alternatives for Obesity Hypoventilation Syndrome. Pickwick Study. Am J Respir Crit Care Med. 2015 Jul 1;192(1):86-95. doi: 10.1164/rccm.201410-1900OC. PMID 25915102